CLINICAL TRIAL: NCT02598167
Title: Assessing Patients Preferences Towards Disease-modifying Therapeutic Options in Relapsing Remitting Multiple Sclerosis
Brief Title: Participants Preferences to Disease Modifying Agents in Relapsing Remitting Multiple Sclerosis Condition
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29715
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- RRMS Population: Participants with a diagnosis of RRMS and being prescribed with a DMT for a period of at least 3 months according to standard local clinical practice will be included.

SUMMARY:
This multi-center non-interventional, observational, cross-sectional study in adult participants with relapsing remitting multiple sclerosis (RRMS) will evaluate the participants' preferences for disease modifying treatments (DMT) in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged greater than or equal to (>/=) 18 years
* Participants who have a diagnosis of RRMS as documented in their medical records
* Participants who have been prescribed a DMT for at least 3 months
* Participants who have an expanded disability status scale (EDSS) score of 1-6 points

Exclusion Criteria:

- Participants with any personal or medical condition that in opinion of the investigator would interfere with or make impossible proper participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of RRMS and being prescribed with a DMT for a period of at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-02-23 (Actual); Study Completion 2016-02-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Serious Adverse Events (Severe Life-Threatening or Less Severe) | Up to 3 months
Percentage of Participants With DMT Administration Schedule Preferences | Up to 3 months
Percentage of Participants With DMT Route of Administration Preferences | Up to 3 months
DMT Efficacy Based on Annualized Relapse Rate | Up to 3 months

SECONDARY OUTCOMES:
Participants Education Level | Baseline
Participants Employment Status | Baseline
Participants RRMS Disease Duration | Baseline
Number of Relapses of RRMS in Last 2 Years | Baseline
Duration since Last Relapse of RRMS | Baseline
Participants Current DMT for RRMS | Baseline
Number of Previous DMTs Taken Prior to Switch to Current DMT | Baseline
Expanded Disability Status Scale (EDSS) Score | Up to 3 months
Health-Related Quality of Life Assessment Using Euro-Quality of Life 5 Dimension Questionnaire (EQ-5D) Scale Score | Up to 3 months
Participant's Role in Decision Making measured by the Shared Decision Making Questionnaire 9-item version (SDM-Q-9) Score | Up to 3 months
Cognitive performance as measured by the Medical Outcomes Study Cognitive Functioning Scale (MOS Cog-R) Score | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Spain (18):
  - Hospital Sant Joan Despi Moises Broggi; Servicio de Neurología, Sant Joan Despí, Barcelona
  - Hospital Universitario Marques de Valdecilla; Servicio de Neurología, Santander, Cantabria
  - Hospital General de Castellon; Servicio de Neurología, Castellon, Castellon
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Neurología, Lleida, Lerida
  - Hospital Universitario del Sureste; Servicio de Neurologia, Arganda, Madrid
  - Hospital Universitario Rey Juan Carlos de Móstoles; Servicio de Neurología, Móstoles, Madrid
  - Hospital Quiron de Madrid; Servicio de Neurologia, Pozuelo de Alarcón, Madrid
  - Complejo Hospitalario Universitario de Vigo - Xeral Cies; Servicio de Neurologia, Vigo, Pontevedra
  - Hospital Universitario de Canarias; Servicio de Neurologia, San Cristóbal de La Laguna, Tenerife
  - Hospital del Mar; Servicio de Neurologia, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Neurologia, Córdoba
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Neurologia, Girona
  - Hospital General Universitario Gregorio Marañon; Servicio de Neurologia, Madrid
  - Fundacion Jimenez Diaz; Servicio de Neurología, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Neurologia, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Neurologia, Valencia
  - Hospital Universitario Dr. Peset; Servicio de Neurologia, Valencia
  - Hospital Universitario La Fe; Unidad de Esclerosis Multiple, Valencia